CLINICAL TRIAL: NCT04249193
Title: Effect of Blood Transfusions on Intermittent Hypoxic Episodes in Very Low Birth Weight Infants
Brief Title: Pulse Oximetry Measurement and Transfusions
Acronym: POMAT
Status: Completed | Type: Observational
Sponsor: Christiana Care Health Services (Other)
Collaborators: Temple University Hospital (Unknown); University of Pennsylvania (Other); Pennsylvania Hospital (Unknown)
Responsible Party: Principal Investigator, Kelley Kovatis, Attending Neonatologist, Christiana Care Health Services
Other Study IDs: DDD603862
Record Dates: First submitted 2020-01-24; First posted 2020-01-30 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Hypoxia Neonatal; Premature; Blood Transfusion
Keywords: Transfusion; Intermittent hypoxia
MeSH Terms: conditions — Asphyxia Neonatorum; Premature Birth | interventions — Blood Transfusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Transfusion
  Interventions: Other: Transfusion

INTERVENTIONS:
Other: Transfusion — pRBC and non-pRBC transfusions

SUMMARY:
The primary purpose of this observational study was to determine if pRBC transfusions decrease the frequency of intermittent hypoxia events in very low birth weight infants (VLBW) during the first six weeks of life. The impact on non-pRBC transfusions on the frequency of intermittent hypoxia was also assessed.

ELIGIBILITY:
Inclusion Criteria:

* 23+0 to 28+6 weeks gestational age at birth

Exclusion Criteria:

* Infants with life-limiting diagnoses
* Cyanotic heart disease
* In utero fetal transfusion
* Twin to twin transfusion syndrome
* Isoimmune hemolytic disease
* Severe acute hemorrhage
* Acute shock
* Sepsis with coagulopathy
* Need for perioperative transfusion
* Parents opposed to transfusion of blood
* Parents with hemoglobinopathy or congenital anemia

Max Age: 6 Weeks | Sex: All
Age Groups: Child
Study Population: Premature neonates
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Change in number of Intermittent hypoxia | Change in number of intermittent hypoxia before (approximately 8 hours) and after transfusion (approximately 8 hours).
  An intermittent hypoxemia event is defined as a fall in oxygen saturations to less than 80% for >/= 10 secs and <3 minutes with a minimal time interval of 4 seconds between events.

SECONDARY OUTCOMES:
Hypoxia | 8 hours prior to transfusion and 8 hours after transfusion.
  Percent time with oxygen saturations less than 85%, 80% and 75%.

CONTACTS AND LOCATIONS:
Overall Officials: Kelley Z Kovatis, MD, Principal Investigator — Christiana Care Health Services, Inc
Locations (3):
- United States (3):
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No